CLINICAL TRIAL: NCT03049566
Title: Discontinuation of Low-dose Acetylsalicylic Acid Before Elective Non-cardiac Surgery: a Preoperative Monocentric Cross-sectional Study
Brief Title: Low-dose Acetylsalicylic Acid Before Non-cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: WF03013
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Surgery; Platelet Dysfunction
Keywords: Bleeding; Adverse Cardiac Events; Adherence, Medication; Aspirin; Acetylsalicylic acid
MeSH Terms: conditions — Hemorrhage; Cardiovascular Diseases; Medication Adherence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- preoperative questionnaires: Patients on long-term acetylsalicylic acid undergoing non-cardiac surgery
  Interventions: Other: preoperative questionnaires

INTERVENTIONS:
Other: preoperative questionnaires — no intervention, cross-sectional survey in a single group

SUMMARY:
This study aims to assess independent factors associated with the clinical decision to discontinue ASA preoperatively in patients undergoing elective non-cardiac surgery.

DETAILED DESCRIPTION:
Acetylsalicylic acid (ASA) is widely used for primary and secondary prevention of cardiovascular diseases. A prothrombotic rebound phenomenon after aspirin cessation has been reported. ASA withdrawal is associated with an increased incidence of adverse cardiac events. In individuals with previous percutaneous coronary intervention (PCI), cessation of ASA may cause stent thrombosis or myocardial infarction. However, many patients undergo non-cardiac surgery within the first two years after PCI. Perioperatively, two counteracting risks have to be taken into account, first, the risk of thromboembolic complications, if ASA medication is discontinued and second, the risk of surgical bleeding, if ASA therapy is continued. However, factors contributing to preoperative decision-making for ASA-withdrawal are still unclear.

This study aims to assess independent factors associated with the clinical decision to discontinue ASA preoperatively in patients undergoing elective non-cardiac surgery. In particular this study aims to determine if the presence of coronary stents is independently associated with ASA discontinuation. Furthermore this study assesses, if benefit-risk-estimates (numerical rating scales) of the patients and the supervising physicians are associated with the decision to withdraw ASA.

Study design

Patients on long-term ASA undergoing non-cardiac surgery as well as their supervising anesthesiologist participate in a preoperative survey. Detailed information about ASA medication, perioperative ASA use, comorbidities, factors that might be associated with the decision to discontinue ASA preoperatively and benefit-risk-estimates (numerical rating scales) are sampled by questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years and older
* Scheduled for elective non-cardiac surgery
* Regular long-term ASA use, defined as daily low-dose (≤100mg) ASA therapy, even if ASA-medication was interrupted within the last 30 days before study inclusion

Exclusion Criteria:

* < 18 Years
* No consent given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective non-cardiac surgery, who present in the pre-assessment clinic of the University Medical Center Hamburg-Eppendorf during the study recruitment period, are screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 805 (Actual)
Dates: Start 2014-02-10 (Actual); Primary Completion 2014-12-30 (Actual); Study Completion 2014-12-30 (Actual)

PRIMARY OUTCOMES:
Preoperative discontinuation of acetylsalicylic acid medication | 1 day
  questionnaires (cross-sectional observation during preoperative assessment)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Zöllner, Professor, Study Director — Department of Anesthesiology, Center of Anesthesiology and Intensive Care Medicine, University Medical Center Hamburg-Eppendorf; Martin Petzoldt, Dr. med., Principal Investigator — Department of Anesthesiology, Center of Anesthesiology and Intensive Care Medicine, University Medical Center Hamburg-Eppendorf
Locations (1):
- Department of Anesthesiology, Center of Anesthesiology and Intensive Care Medicine, University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No